CLINICAL TRIAL: NCT01286064
Title: Role of Natural Fluorescence of Human Blood Plasma in Patients With Colorectal Cancer.
Brief Title: Colorectal Cancer Detection by Means of Optical Fluoroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Alberto Vannelli, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: INT-D178768
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2010-09

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma,; colorectal tumors,; endogenous porphyrins,; fluorescence,; tumor markers.
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient with colo-rectal cancer (Experimental): fluorescence spectra will be mainly characterized by the presence of an emission peaking at 620-630 nm
  Interventions: Device: Optical Fluoroscopy
- patient without colo-rectal cancer (Active Comparator): fluorescence spectra will be characterized by the absence of an emission peaking at 620-630 nm
  Interventions: Device: Optical Fluoroscopy

INTERVENTIONS:
Device: Optical Fluoroscopy — Lithium-heparin was added to the blood samples to prevent coagulation. The samples were then centrifuged and the plasma was removed without disturbing the buffy coat and the erythrocyte sediments. The separated changes in the enzyme associated with heme biosynthesis have been reported for peripheral mononuclear cells in patients with epithelial tumors and metastatic spread. plasma was stored at -20 °C until assayed. For fluorescence measurements, analytical grade acetone was added to plasma in a 1:1 ratio by volume and the mixture was centrifuged. The clear supernatant was placed in a quartz cuvette of 1 cm path length for further analysis. Fluorescence analysis of blood plasma was performed by means of a spectrofluorometer (Model F-3000, Hitachi, Ltd., Tokyo, Japan).
  Arms: patient with colo-rectal cancer
Device: Optical Fluoroscopy — Lithium-heparin was added to the blood samples to prevent coagulation. The samples were then centrifuged and the plasma was removed without disturbing the buffy coat and the erythrocyte sediments. The separated changes in the enzyme associated with heme biosynthesis have been reported for peripheral mononuclear cells in patients with epithelial tumors and metastatic spread. plasma was stored at -20 °C until assayed. For fluorescence measurements, analytical grade acetone was added to plasma in a 1:1 ratio by volume and the mixture was centrifuged. The clear supernatant was placed in a quartz cuvette of 1 cm path length for further analysis. Fluorescence analysis of blood plasma was performed by means of a spectrofluorometer (Model F-3000, Hitachi, Ltd., Tokyo, Japan).
  Arms: patient without colo-rectal cancer

SUMMARY:
The aim of the present prospective study was to investigate the fluorescence emission of human blood plasma of patients with colorectal cancer.

For years, serum tumor markers have been studied for the diagnosis and follow-up of colorectal cancer, among which carcinoembryonic antigen (CEA) has achieved promising results. However, the sensitivity of CEA for colorectal cancer is less than 25% and elevated CEA levels also occur in patients with benign disease, as well as in patients with other carcinomas. Nevertheless, surveillance programs are often based on the CEA test and combination with other markers is at present a matter of research. Alternative methods based on optical fluoroscopy have been introduced in experimental stages for clinical diagnosis of cancer. Few studies have been reported on the application of native fluorescence spectroscopy of biofluids in the diagnosis of tumoral diseases. The above reported findings prompted us to investigate the fluorescence emission of human blood plasma of patients with colorectal cancer. For this purpose, the blood of patients was collected and the fluorescence Preliminary measurements on plasma of patients bearing colon cancer showed that the fluorescence spectra were mainly characterized by the presence of an emission peaking at 620-630 nm, whose excitation spectrum peaked at 405 nm. Hence, an excitation wavelength of 405 nm was selected for the study. The fluorescence emission spectra were recorded in the range of 430-700 nm.

DETAILED DESCRIPTION:
Eligibility criteria: Gastrointestinal disease or clinical symptoms related to colorectal cancer risk submitted to endoscopy. Exclusion criteria consisted of age younger than 18 years, history of psychiatric illness, and preoperative radiotherapy.

Outcome: investigated the possible role of the native fluorescence of blood plasma in the management of colorectal cancer (CRC) and its feasibility as a new tumor marker. Sample of blood was collected from asymptomatic blood donors and from CRC patients. The native fluorescence of blood plasma was measured using a conventional spectrofluorimeter.

ELIGIBILITY:
Inclusion Criteria:

Gastrointestinal disease clinical symptoms related to colorectal cancer risk endoscopy

Exclusion Criteria:

Age younger than 18 years or more than 75 years, history of psychiatric illness, preoperative chemo/radiotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer detection by means of optical fluoroscopy | 18 months
  investigated the possible role of the native fluorescence of blood plasma in the management of colorectal cancer (CRC) and its feasibility as a new tumor marker.

CONTACTS AND LOCATIONS:
Overall Officials: alberto vannelli, md, Study Director — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy, Italy

REFERENCES:
- See also: Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy — http://www.istitutotumori.mi.it/